CLINICAL TRIAL: NCT03440749
Title: Rhythm and the Multisensoriality's Effects on the Motor Development in Children With Cerebral Palsy
Brief Title: Rhythm and Multisensoriality's Effects on the Motor Development in Children With Cerebral Palsy
Acronym: APP-PaC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/17/0158; 2017-A01969-44 (Other: Toulouse Hospital)
Record Dates: First submitted 2018-02-13; First posted 2018-02-22 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy
Keywords: rhythm; serial Reaction Time Task
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Comparative monocentric physiopathological study with 2 groups of children : children with cerebral palsy and children age-matched for the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children with Cerebral Palsy (PC) (Experimental): Serial reaction time task: repeating a sequence of movements according to the luminous stimuli
  Interventions: Other: luminous stimuli
- Control Group (Active Comparator): Serial reaction time task: of movements according to the luminous stimuli
  Interventions: Other: luminous stimuli

INTERVENTIONS:
Other: luminous stimuli — The child is placed in front of a screen on which 4 luminous stimuli are presented on a horizontal plane. Four buzzers are placed in front of him, each buzzer corresponds to the position of a stimulus. Child had to push the buzzer corresponding to the place of the luminous stimuli.
  Other Names: Serial reaction time task

SUMMARY:
Cerebral palsy (CP) affects the motor function but also the cognitive function of the child. Physical activity brings motor and cognitive benefits and appears as an important aspect of the therapy that is offered to them.

The child is seating in front of a computer, seating comfortably on a chair during 1 hour. The experimental task consists in learning a sequence of taps on "Serial reaction time task" type buzzers (SRTT) in which the child must press a buzzer corresponding to one of the 4 squares that on the screen. The sequence corresponds to 10 steps in a particular order.

DETAILED DESCRIPTION:
Cerebral palsy (CP) affects the motor function but also the cognitive function of the child. Physical activity brings motor and cognitive benefits and appears as an important aspect of the therapy that is offered to them. In particular, the learning of movements in the presence of multisensory rhythmic information seems to have beneficial effects at the cognitive and motor level. The present study aims to test the respective effects of rhythm and multisensoriality on motor learning in children with cerebral palsy.

The motor learning task is known as the "Serial Reaction Time Task" (SRTT). It consists in repeating a sequence of movements of the upper limbs using visual-spatial information alone (V). It will test the addition of synchronous auditory stimulation to visual information or rhythmic auditory stimulation(VAR), to contrast with a control condition with non-rhythmic auditory stimulation (VANR). The performance of the children will be measured by the reaction time (RT), its stability and the number of errors made throughout the motor learning.

The child is placed in front of a screen on which 4 luminous stimuli are presented on a horizontal plane. Four buzzers are placed in front of him, each buzzer corresponds to the position of a stimulus. The stimuli light up in a predetermined sequence (10 positions) and the child must press the buzzer corresponding to the position of the stimulus that comes on. Four blocks of 5 sequences are repeated to test the general learning (B1 to B4) and then a block of random stimuli is presented to test the specific learning of the sequence (B5).

ELIGIBILITY:
Inclusion Criteria:

For all children:

* Age between 6 and 14 years
* Obtaining the informed consent of the person possessing parental authority for all children

For children with Cerebral Palsy:

* Diagnosis of spastic cerebral palsy of levels GMFCS I to IV
* Ability to press buzzers with the palm of the hand, Manual Ability Classification System (MASC) I to IV
* Ability to understand instructions ("tap a buzzer along with a picture or sound") (investigator's appreciation)

For control children: no pathology diagnosed

Exclusion Criteria:

For all children:

* Children with a characteristic psychiatric pathology.
* Disorders of the understanding
* Hearing deficiency
* Uncorrected visual impairment

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Time reaction (TR) | 1 hour
  - The TR is the Reaction Time between the appearance of the stimulus and the response. It represents the speed with which the child pressed the key in response to the lighting of the square.

SECONDARY OUTCOMES:
Number of errors | 1 hour
  The number of errors corresponds to pressing a key that does not correspond to the position of the lit square.

OTHER OUTCOMES:
Multisensory integration degree | 1 hour
  Multisensory integration degree evaluated in pre-test
Degree of synchronization | 1 hour
  Degree of synchronization evaluated in pre-test

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Marque, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No